CLINICAL TRIAL: NCT06583512
Title: Invasive Pulmonary Aspergillosis Treatment Duration of Posaconazole-initiated Antifungal Strategy in Patients with Hematological Malignancies: a Prospective, Single-center Study
Brief Title: Treatment Duration of IPA
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Sun Yuqian, Principal Investigator, Peking University People's Hospital
Other Study IDs: 2024PHB035-001
Record Dates: First submitted 2024-08-06; First posted 2024-09-04 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Invasive Aspergillosis; Antifungal Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to identify the duration of posaconazole-initiated antifungal treatment for IPA in patients with hematological malignancies and to explore the value of monitoring immune factors and cells in IPA treatment in order to assess practices in IPA management in Chinese hematology patients including tools to evaluate duration and discontinuation. The main question it aims to answer is:

Does any indicators that could be used to guide the duration of IPA treatment? Does immune factors have value in monitoring IPA treatment? We will not do any interventions to participants. Participants will be monitored routinely for their clinical characteristics, microbiological test( including G/GM Test, Blood culture), Imaging examination, Blood routine, the number and function of immune cells, cytokines(IL-1β/IL-2/IL-4/IL-8/IL-10/IL-12/IL-17/IFN-α/IFN-γ/TNF-α)， and we will collect these datas for analysing.

DETAILED DESCRIPTION:
1. A total of 15 patients will be involved in the study.
2. For each patient, the investigator will first evaluate the patient to determine if the patient meets the enrollment criteria and does not meet any of the exclusion criteria.
3. For the patients included in the study, the investigators will collect their blood RT, immune cell count and function, and cytokine levels (including IL-1β/IL-2/IL-4/IL-5/IL-6/IL-8/IL-10/IL-12/IL-17/INF-γ/INF-α/TNF-α et al).
4. Closely monitor the patient's status and discontinue antifungal therapy if the patient meet the 4 critera: ①PMNs recovery>500；②previous signs/symptoms of active IPA (such as fever) has been resolved; ③nagative mycological evidence; ④CT: the reduction in the size of the lesion must exceed 90% or stable cave. If the patient does not meet any of these criteria, antifungal therapy is continued until the 4 critera are met.
5. Blood RT, neutrophil count and function, and cytokine levels (IL-1β/IL-2/IL-4/IL-5/IL-6/IL-8/IL-10/IL-12/IL-17/INF-γ/INF-α/TNF-α) were collected at the time of stopping antifungal therapy and at 2, 4, 8, and 12 weeks after stopping treatment. At the same time, the patient's symptoms (cough, hemoptysis, fever, etc. )and signs (chest pain, etc. ) were observed and the patient's microbiology examination results (blood G/GM text, fungal culture, etc. ) and imaging examination results (CT, etc.) were collected at the follow-up.
6. Follow-up will be conducted instantly if any symptom, sign, or text result suspected IPA after discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form signed
2. Patient with hematological malignancies
3. Patients with posaconazole-initiated antifungal therapy
4. Treatment duration ≥12w

Exclusion Criteria:

1. Refuse to enroll
2. Pregnancy or breastfeeding women
3. Are expected to survive no more than 72 h
4. Fungal or mycobacterial lung co infection at time of IPA diagnosis
5. Hematological malignancy with lung location
6. Disseminated aspergillosis (lung and sinus aspergillosis can be included)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: These patients had a hematological malignancies, and then had a invasive pulmonary aspergillosis. They were treated by posaconazole as their initiated drug and the treatment duration last for more than 12 weeks.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The duration of posaconazole-initiated antifungal treatment therapy for IPA in patients with hematological malignancies | 12 weeks after discontinuation of posaconazole-initiated antifungal therapy
  The primary outcome is the duration of posaconazole-initiated antifungal treatment therapy for IPA in patients with hematological malignancies

SECONDARY OUTCOMES:
All-cause mortality on 2/4/8 /12 weeks after discontinuation | 12 weeks after discontinuation of posaconazole-initiated antifungal therapy
  The mortality of patients died for any reasons on 2/4/8/12 weeks after discontinuation of antifungal therapy
IFI-free survival rate on 2/4/8/12 weeks after discontinuation | 12 weeks after discontinuation of posaconazole-initiated antifungal therapy
  The IFI-free survival rate of patients on 2/4/8/12 weeks after discontinuation of antifungal therapy
Clinical success rate of posaconazole-initiated antifungal therapy | 12 weeks after discontinuation of posaconazole-initiated antifungal therapy
  The rate of patients who achieved clinical remission after posaconazole-initiated antifungal therapy
The proportion of patients who restarted treatment after discontinuation | 12 weeks after discontinuation of posaconazole-initiated antifungal therapy
  After discontinuation of posaconazole-initiated antifungal therapy ,the rate of patients who restarted treatment of antifungal
Analysis of criteria that could be used to guide the discontinuation of IPA treatment | 12 weeks after discontinuation of posaconazole-initiated antifungal therapy
  After discontinuation of posaconazole-initiated antifungal therapy , the related therapy options will be analyzed and the investigators will do some recommmendations for the discontinuation of IPA treatment.
The value of immune factors (IL-1β/IL-2/IL-4/IL-5/IL-6/IL-8/IL-10/IL-12/IL-17/IFN-α/IFN-γ/TNF-α) and cells (the count of neutrophil and lymphocytes) | from the beginning of posaconazole-initiated treatment to 12 weeks after discontinuation of posaconazole-initiated antifungal therapy
  The blood RT、neutrophil function、lymphocyte count/function 、cytokine (IL-1β/IL-2/IL-4/IL-5/IL-6/IL-8/IL-10/IL-12/IL-17/IFN-α/IFN-γ/TNF-α) will be recorded and analysed at the beginning of the posaconazole-initiated treatment and 2/4/8/12 weeks after discontinuation of treatment.
The trend of immune factors (IL-1β/IL-2/IL-4/IL-5/IL-6/IL-8/IL-10/IL-12/IL-17/IFN-α/IFN-γ/TNF-α) and cells (the count of neutrophil and lymphocytes) | from the beginning of posaconazole-initiated treatment to 12 weeks after discontinuation of posaconazole-initiated antifungal therapy
  The blood RT、neutrophil function、lymphocyte count/function 、cytokine (IL-1β/IL-2/IL-4/IL-5/IL-6/IL-8/IL-10/IL-12/IL-17/IFN-α/IFN-γ/TNF-α) will be recorded and analysed at the beginning of the posaconazole-initiated treatment and 2/4/8/12 weeks after discontinuation of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yuqian Sun, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No